CLINICAL TRIAL: NCT01607060
Title: Impact of Laxative Therapy With Lactulose in the Evolution of Organ Dysfunction in Critically Ill Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo Palácio de Azevedo, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lactulona
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2012-10

CONDITIONS: Constipation
Keywords: Critically ill patients; intestinal failure
MeSH Terms: conditions — Constipation; Intestinal Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactulone (Experimental): Patients receiving lactulone
  Interventions: Drug: Lactulone
- Control (Active Comparator): Observational group. Compare to lactulone group.
  Interventions: Drug: Lactulone

INTERVENTIONS:
Drug: Lactulone — Patients will receive lactulone to daily laxation

SUMMARY:
MAIN FEATURES OF THE STUDY: therapeutic intervention. Constipation is a frequent complication in critical ill patients. The disaccharide lactulose has a laxative osmotic activity. Given the scant evidence and the potential risk associated with constipation in seriously ill patients, this study aims to assess the impact of laxative therapy in the prognosis of critically ill patients.

Study hypothesis: Constipation is part of the clinical spectrum of intestinal dysfunction and if treated can result in improved prognosis for critically ill patients.

DETAILED DESCRIPTION:
OBJECTIVES: Evaluate the impact of daily laxative therapy in the prognosis of critically ill patients through the evaluation of organ failure by the sequential organ failure score assessment (SOFA). Will also be evaluated morbidity data, namely incidence of bloodstream infection, pneumonia and severe sepsis, days free of mechanical ventilation, length of hospital stay, ICU and hospital mortality.

The study will be conducted in two intensive care units of Hospital Sao Paulo, UNIFESP. Inclusion criteria: patients who are mechanically ventilated, with prediction to stay in the ICU for more than three days and getting at least 20% of full nutritional support in the form of enteral nutrition. Patients will be randomized into two groups: Group 1 - patients treated according to medical prescription. Group 2 - patients will receive lactulone in order to evacuate daily. The patient included in the intervention group will receive latulose 30 ml of 8 in 8 hours. Patients will be monitored, adjusted doses and procedures, if necessary. It is intended to include 44 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients expected to stay for 3 more days, on mechanical ventilation and receiving at least 20% of calculated nutrient intake enterally.

Exclusion Criteria:

* younger than 18 years,
* pregnancy,
* contraindication to enteral nutrition,
* patients with liver disease,
* contraindications to the use of lactulose,
* patients with poor prognosis or without full therapeutic indication investment,
* presence of colostomy or ileostomy,
* intestinal diseases,
* such as disease Crohn's,
* ulcerative colitis,
* short bowel syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change in SOFA score | At the moment of inclusion and 14 days latter
  Will evaluate the change in SOFA score between the time of enrollment and 14 days after enrollment, or discharge, or death if it occurs before that date.

CONTACTS AND LOCATIONS:
Locations (1):
- São Paulo Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Azevedo RP, Freitas FG, Ferreira EM, Pontes de Azevedo LC, Machado FR. Daily laxative therapy reduces organ dysfunction in mechanically ventilated patients: a phase II randomized controlled trial. Crit Care. 2015 Sep 16;19(1):329. doi: 10.1186/s13054-015-1047-x. PMID 26373705